CLINICAL TRIAL: NCT02860455
Title: Role of Pulse Co-oximetry in Prehospital Emergency Medical Service Management of Suspected Carbon Monoxide Poisoning : A Prospective Multicenter Study.
Brief Title: Role of Pulse Co-oximetry for Detecting Carbon Monoxide Poisoning in the Prehospital Emergency Medical Service Setting
Acronym: CO-OX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: French Society of Emergency Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8869
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Carbon Monoxide Poisoning
Keywords: CO poisoning; CO-oximetry; Pulse oximetry; Carbon monoxide saturation (SpCO); Emergency Department; Sensitivity; Specificity
MeSH Terms: conditions — Carbon Monoxide Poisoning; Emergencies; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SpCO and COHb measurement (Other): SpCO measurement (Experimental) : Non invasive pulse CO-oximetry will be carried out in all patients simultaneously with venous blood sampling for standard laboratory blood gas analysis, at time of prehospital management by emergency medical services
  COHb measurement (Active comparator) : Blood carboxyhemoglobin testing will be carried out in all patients
  Interventions: Device: RAD57 measurement (SpCO); Device: CO-oximeter

INTERVENTIONS:
Device: RAD57 measurement (SpCO) — SpCO measurement (Experimental)
  Non invasive pulse CO-oximetry will be carried out by prehospital emergency nursing staff trained in the use of the Rad-57 pulse CO-oximeter (Masimo, Inc., Irvine, CA, USA), using the adult sized sensor (Sensor, Rev. B) placed on the 3rd or 4th digit, according to manufacturer recommendations. Nail polish will be removed if necessary. SpCO was expressed in total percentage of hemoglobin.
  Other Names: Non invasive pulse CO-oximetry
Device: CO-oximeter — COHb measurement (Active Comparator)
  Venous blood will be collected into EDTA treated tubes (Beckton Dickinson) prehospitally and sent to the toxicology laboratory for further carboxyhemoglobin testing. Blood carboxyhemoglobin will be analyzed by derivative spectrophotometry using an automated CO-oximeter (IL 682, Instrumentation Laboratory SpA V.le Monza 338-20128 Milan, Italy). Blood carboxyhemoglobin will be detected within a range of 0-100% and accuracy of 0.5% and reported as percentage of total haemoglobin.

SUMMARY:
The RAD-57 pulse CO-oximeter is a lightweight device allowing non-invasive measurement of blood carboxyhemoglobin. Previous studies comparing RAD-57 measurements (SpCO) to standard laboratory blood gas analysis (COHb) have reported contradictory results.

the RAD-57 pulse CO-oximeter could be useful as a first-line screening test for acute CO poisoning, enabling rapid detection and management of patients with suspected CO poisoning in the prehospital emergency setting This study assesses the diagnostic value of pulse CO-oximetry, comparing SpCO to standard laboratory blood measurement for prehospital management of patients with suspected carbon monoxide (CO) poisoning.

DETAILED DESCRIPTION:
Transcutaneous SpCO will be obtained using the RAD-57 simultaneously with blood sampling for laboratory blood gas analysis, at the time of prehospital management by emergency medical services. The diagnostic performance of SpCO for the screening of CO poisoning will be determined using ROC curve analysis, and Blood COHb levels >5% and 10% as the reference standard for CO poisonning for non-smokers and smokers respectively. Correlation between SpCO and COHb will be assessed using Bland and Altman's method.

ELIGIBILITY:
Inclusion criteria:

* Patient aged 18 years or older
* Patient managed by prehospital emergency medical services.
* Patient with a suspected CO exposure presenting or not with clinical signs of CO poisoning

Exclusion criteria:

* Patient for whom venous blood sampling cannot be obtained prehospitally
* Patient for whom SpCo measurement cannot be performed prehospitally (cardiac arrest, peripheral vasoconstriction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2012-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
SpCO optimal threshold value for detection of CO poisoning | Baseline
  prehospital medical management

SECONDARY OUTCOMES:
SpCO level | Baseline
  prehospital medical management
COHb Blood carboxyhemoglobin level | Baseline
  prehospital medical management

CONTACTS AND LOCATIONS:
Overall Officials: Mustapha Sebbane, MD, PhD, Principal Investigator — Montpellier University hospital - Emergency department
Locations (1):
- Montpellier University hospital - Emergency department, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided